CLINICAL TRIAL: NCT01189838
Title: The Expression and Effect of Cyr61 in Urinary Tract Transitional Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Other Study IDs: 098055-3
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-01

CONDITIONS: Carcinoma, Transitional Cell
Keywords: Cancer; cysteine-rich 61; prognosis; transitional cell carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Surgical resection of tumor
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low Cyr61: Low Cyr61 immunohistochemical stain in patients' TCC tumor
- High Cyr61: High Cyr61 immunohistochemical stain in patients' TCC tumor

SUMMARY:
Cysteine-rich 61 (Cyr61), a member of "CCN" family, regulates cell migration, proliferation, apoptosis, and angiogenesis, cell adhesion, migration, proliferation, survival, differentiation, apoptosis, angiogenesis, and extracellular matrix production. Evidences show strong correlations of aberrant Cyr61 expression in cancers of numerous organs and tissues. However, the expression and effect of Cyr61 in transitional cell carcinoma (TCC), the most common urinary tract cancer in Taiwan, remains undiscovered. Based on previous studies of Cyr61 in other cancer, the investigators hypothesize that Cyr61 may mediate TCC cell proliferation and migration; and associated with disease progression and recurrent. Thus the investigators conduct this project to study the role of Cyr61 in the pathogenesis of TCC. The investigators will retrospectively review medical history of patients with TCC treated at our institutes. Cyr61 immunohistochemical stain of their surgical samples will be performed. The correlation of Cyr61 expression of TCC and patients' clinical courses will be investigated.

DETAILED DESCRIPTION:
1. Patients: as shown in inclusion criteria
2. Surgical samples Surgical specimens from included patients with TCC who underwent surgery will be collected. The samples will be examined histologically for the presence of tumor cells. Independent pathologists who are blinded to the records of the patients will perform histological examinations. Tumor grade is determined on the basis of cytological features. There are three grades of TCC, as proposed by Mostofi et al. and adopted by the American Bladder Tumor Registry of the World Health Organization. These are based on degree of anaplasia: Grade 1 tumors show mild cytological atypia and rare mitosis; Grade 2 tumors show moderate cytological atypical and the presence of mitotic figures; and Grade 3 tumors show severe cytological atypia and frequent mitotic figures. Lymph node metastasis, lymphatic invasion, and venous invasion will be evaluated by pathology reports and image study. Clinical staging of TCC is based on the American Joint Committee on Cancer staging (AJCC) TNM system.
3. Immunohistochemical stain Paraffin-embedded, formalin-fixed surgical specimens were collected for Cyr61 immunohistochemical staining. Heat-induced epitope retrieval will be performed with a pressure cooker and TRIS buffer (pH 9.0) for 2 min. They will be allowed to cool for 15 min, rinsed in distilled water twice and in PBS for 5 min. The sections will then be treated with 0.5% hydrogen peroxidase/PBS for 20 min at room temperature to block the endogenous peroxidase. They will subsequently be blocked with 10% normal goat serum for 30 min at room temperature, and then incubated with polyclonal anti-Cyr61 antibody (Santa Cruz, CA) at 4°C overnight. The specific antibodies will be omitted in sections as negative controls. The sections will be washed three times in PBS/0.2% Triton X-100 for 10 min and incubated with biotin-conjugated secondary antibodies (DAKO, Carpinteria, CA) for 1 hour at room temperature the following day. They will then be incubated with the avidin-biotin-peroxidase reagent (DAKO) for another 1 hour at room temperature. After three washes in PBS/0.2% Triton X-100 for 10 min each, the reactions on sections will be detected with peroxidase substrate containing diaminobenzidine chromagen (DAKO). The slides will be counterstained with hematoxylin. If >50% of the tumor cells are positively stained, the specimen will be grouped as "positive". All other staining results will be regarded as negative.
4. Statistical analysis For statistical analysis, P values are based on two-sided, parametric Student's t tests. A P value of <0.05 on the basis of at least three independent sets of experiments is considered to be statistically significant. In the clinical sets of project, Chi-squire test and Student's t test will be used to study the association of Cyr61 expression with single clinical factors (age, gender, pathology, and grade). Kaplan-Meier survival curves for patients with positive versus negative Cyr61 expression will be plotted and log-rank test will be used for comparing the equality of the two survival curves. Cox proportional hazard model will also be developed to correlate the clinical characteristics, survival, and the expression of Cyr61.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age>18 years) with TCC who received surgery at Far Eastern Memorial Hospital and National Taiwan University Hospital from 2004 to 2008.

Exclusion Criteria:

* Refuse to participate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will retrospectively review adult patients (age>18 years) with TCC who received surgery at Far Eastern Memorial Hospital and National Taiwan University Hospital from 2004 to 2008.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Fu Lai, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan